CLINICAL TRIAL: NCT06701591
Title: Efficacy of Combined Kinesio-Taping With Chest Physiotherapy Program on Pain, Pulmonary Function, Respiratory Muscle Strength and Quality of Life After Mastectomy: A Randomized Controlled Trial
Brief Title: Kinesio-Taping and Chest Physiotherapy Program After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 6905
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-12

CONDITIONS: Mastectomy
Keywords: kinesiotaping; pain; physiotherapy; pulmonary function; respiratory muscle strength; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Kinesiotaping group) (Experimental): Participants will be seated on a chair, KT will be applied bilaterally at the end of the expiration on the fifth to sixth and ninth to tenth intercostal muscles transversally and on the anterior and posterior axillary line longitudinally with 50% tension. In order to stimulate the muscle and support the function, the stimulation technique is usually applied from the origin to the insertion of the muscle with the recommended stretching of 25 to 50%.
  Additionally, traditional physical therapy program will be conducted to participants in the study group.
  Interventions: Other: Kinesiotaping; Other: chest physical therapy
- Group B (control group) (Active Comparator): They will receive the chest physical therapy program which is consisted of deep breathing exercises, postural drainage, cough, 3 times /week for 4 weeks.
  Interventions: Other: chest physical therapy

INTERVENTIONS:
Other: Kinesiotaping — Participants will be seated on a chair, KT will be applied bilaterally at the end of the expiration on the fifth to sixth and ninth to tenth intercostal muscles transversally and on the anterior and posterior axillary line longitudinally with 50% tension. In order to stimulate the muscle and support the function, the stimulation technique is usually applied from the origin to the insertion of the muscle with the recommended stretching of 25 to 50%.
  Arms: Group A (Kinesiotaping group)
Other: chest physical therapy — The chest physical therapy program is consisted of deep breathing exercises, postural drainage, and cough.

SUMMARY:
The modified radical mastectomy (MRM) is a major surgical approach that necessitates the dissection of axillary lymph nodes. As a result, there is more bleeding and the treatment takes longer time. This treatment is used to treat locally advanced breast cancer. Numerous factors, including pain and respiratory depression from general anaesthesia, can impair respiratory function during the post-operative period. Pain causes the thoracic cage's post-operative movement to be restricted and the breathing muscles to become inhibited.

DETAILED DESCRIPTION:
KT is a new technology that is being used in the treatment of post-surgical and respiratory problems, among other innovative evidence-based therapeutic options in patient care. Recently, this method is useful for treating a variety of sports-related and musculoskeletal disorders, as well as pain management. According to a small body of research on the usefulness and efficacy of KT in treating respiratory conditions in patients with chronic obstructive pulmonary disease (COPD), it can lead to improvements in respiratory muscle strength and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 30 and 50 years
* Participants after modified radical mastectomy
* Participants able to comprehend instructions.
* Cooperative participants, and willing to participate in the study.

Exclusion Criteria:

* Participants having sensitive skin, scars, or lesions.
* Participants with unhealed incisions at the site of application.
* Participants with uncontrolled diabetes.
* Participants with deep vein thrombosis.
* Participants with previous chest diseases.
* Pregnancy.
* Participants with altered sensations.
* Participants with allodynia.
* Participants with active infection.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 4 weeks
  The visual representation of the pain range that a patient thinks they might experience is called a linear scale. The score is ranged from 0 to 10. The least the score, the better results. While, the higher the score, the worst the results.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 4 weeks
  The forced vital capacity (FVC) will be measured by spirometer.
forced expiratory volume at first second (FEV1) | 4 weeks
  forced expiratory volume at first second (FEV1) will be measured by spirometer.
Forced expiratory volume at first second /Forced vital capacity ratio. | 4 weeks
  Forced expiratory volume at first second /Forced vital capacity ratio will be measured by spirometer.
Respiratory muscle strength | 4 weeks
  Respiratory muscle strength will be measured by assessing the maximal inspiratory and maximal expiratory pressures (MIP) and maximal expiratory pressures (MEP).
Quality of life | 4 weeks
  Quality of life will be measured by the Short Form-36 (SF-36). It is a questionnaire with eight subscales that gives information about the health status and quality of life of the person. Scores on each subscale range from 0 to 100, with 0 corresponding to the worst health status and 100 to the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Director — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months after publication

REFERENCES:
- [Derived] Elsherbini DMA, Eladl HM, Allam NM, Abulfaraj M, El-Sherbiny M, Nosseir N, Maghrabi A, Jamal W, Abdelrahman MMA, Eladl MA. Efficacy of combined Kinesio-taping with chest physiotherapy program on pain, pulmonary function, respiratory muscle strength and quality of life after mastectomy: a randomized controlled trial. Front Med (Lausanne). 2026 Jan 22;12:1664210. doi: 10.3389/fmed.2025.1664210. eCollection 2025. PMID 41657582